CLINICAL TRIAL: NCT02662036
Title: A Prospective Trial to Assess Analgesic Efficacy of Liposomal Bupivacaine vs. Bupivacaine HCL as a Tap Block After Abdominally Based Autologous Breast Reconstruction
Brief Title: Analgesic Efficacy of Liposomal Bupivacaine vs. Bupivacaine HCL as a Tap Block After Abdominally Based Autologous Breast Reconstruction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis showed that there was no difference between the two drugs
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201601064
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Mammaplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Bupivicaine (Active Comparator): -TAP block of 30 cc of 0.25% bupivicaine
  Interventions: Drug: Bupivicaine HCL
- Group 2: Liposomal bupivacaine (Experimental): -TAP block of 266 mg/30 cc liposomal bupivacaine
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Bupivicaine HCL
  Other Names: Bupivicaine
  Arms: Group 1: Bupivicaine
Drug: Liposomal bupivacaine
  Other Names: Exparel
  Arms: Group 2: Liposomal bupivacaine

SUMMARY:
This study will evaluate the efficacy of analgesia provided by liposomal bupivacaine (Exparel) when compared to bupivacaine HCL as a transverse abdominis plane (TAP) block in terms of discharge milestones, opioid use, costs, and patient-reported satisfaction at 12, 24, and 72 hours. The investigators propose that Exparel will lower opioid use, length of stay, and overall cost of abdominally-based autologous breast reconstruction, and will lead to greater patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for abdominal-based autologous breast reconstruction (DIEP, MS-TRAM, or TRAM).
* At least 18 years of age.
* Female.
* Able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Cognitive impairment.
* History of abdominal surgery precluding free flap donor site.
* Allergy or intolerance to bupivacaine or "amide" anesthetics.
* Significant preoperative chronic pain (requiring daily narcotics) or neuropathic pain (requiring daily use of pregabalin or gabapentin) within the previous 3 months.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Myckatyn, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Started | 35 | 35
Completed | 22 | 22
Not Completed | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Median (Full Range); unit: years] | 51 [27 to 78] | 47 [34 to 67] | 48.5 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 32 | 34 | 66
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 30 | 28 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Baseline QoR [Median (Full Range); unit: score on a scale] — * Quality of Recovery -15 questionnaire
  * Part A has 10 questions that asks how the participant has been feeling in the last 24 hours with answers ranging from 0=none of the time to 10=all of the time
  * Part B has 5 questions asking the participant if they have had any of the following including pain, nausea, vomiting, anxiety, and depression) with answers ranging from 0=none of the time to 10=all of the time.
  * The total score allowed is 150 (range 0-150) with the higher the number the worse the participant is feeling and the lower the number the better the participant is feeling Population: 10 patients had their surgeries scheduled after the trial closed, 8 were deemed ineligible because they were later found to take preoperative narcotics daily, deviated significantly from the enhanced recovery protocol, or developed recurrent disease prior to surgery. 4 patients withdrew consent and another 4 had missing data.
  score on a scale
    number analyzed (Participants) | 22 | 22 | 44
    (all) | 134 [98 to 147] | 140 [122 to 150] | 136 [98 to 150]

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Opioid Use During Hospital Stay
Time Frame: Up to day of discharge from hospital (expected hospital stay of 5 days)
Measure: Median (Full Range); unit: mg
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
mg
  Intraoperative | 99.5 [15 to 220] | 110.0 [42 to 215]
  Postoperative acute care unit | 0 [0 to 45] | 10 [0 to 100]
  Postoperative floor | 165 [25 to 570] | 138.8 [37.5 to 470]
  Total | 300 [108 to 684] | 283 [90 to 765]
Statistical Analysis 1: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Statistical analysis #1 is for intraoperative opioid use; Test type: Superiority; p = 0.76, Mann Whitney U Test
Statistical Analysis 2: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Statistical analysis #2 is for postoperative acute care unit opioid use; Test type: Superiority; p = 0.38, Mann Whitney U Test
Statistical Analysis 3: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Statistical analysis #3 is for postoperative floor opioid use; Test type: Superiority; p = 0.69, Mann Whitney U Test
Statistical Analysis 4: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Statistical analysis #4 is for total opioid use; Test type: Superiority; p = 0.98, Mann Whitney U Test

2. Secondary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Antiemetic Use During the Hospital Stay
Time Frame: Up to day of discharge from hospital (expected hospital stay of 5 days)
Measure: Median (Full Range); unit: mg
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
mg
  Postoperative acute care unit | 0 [0 to 2] | 0 [0 to 1]
  Floor | 1 [0 to 6] | 1 [0 to 13]
  Total | 1 [0 to 8] | 1 [0 to 13]
Statistical Analysis 1: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Statistical analysis #1 is for postoperative acute care unit antiemetic use; Test type: Superiority; p = 0.28, Mann Whitney U Test
Statistical Analysis 2: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Statistical analysis #2 is for floor antiemetic use; Test type: Superiority; p = 0.62, Mann Whitney U Test
Statistical Analysis 3: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Statistical analysis #3 is for total antiemetic use; Test type: Superiority; p = 0.50, Mann Whitney U Test

3. Secondary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Length of Hospital Stay
Time Frame: Up to day of discharge from hospital, up to 7 days
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
days | 3.56 [2.64 to 4.84] | 2.91 [1.92 to 6.74]
Statistical Analysis 1: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Test type: Superiority; p = 0.20, Mann Whitney U Test

4. Secondary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Time Until Ambulation
Time Frame: Up to 2 weeks post-operation
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
days | 2.20 [0.90 to 3.72] | 1.81 [1.09 to 3.67]
Statistical Analysis 1: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Test type: Superiority; p = 0.64, Mann Whitney U Test

5. Secondary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Duration of Urinary Catheter
Time Frame: Up to 2 weeks post-operation
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
days | 1.27 [0.75 to 3.68] | 1.02 [0.14 to 5.55]
Statistical Analysis 1: Comparison: Group 1: Bupivicaine vs Group 2: Liposomal Bupivacaine; Test type: Superiority; p = 0.38, Mann Whitney U Test

6. Secondary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Pain Scores
Description: * Pain scale uses Wong-Baker FACES Pain Rating Scale
  * The scale uses cartoon faces ranging from 0-10 with 0 meaning no pain and 10 meaning worst possible pain
Time Frame: 12 hours after surgery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
score on a scale | 2.0 [0 to 9] | 0 [0 to 8]

7. Secondary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Pain Scores
Description: as for outcome 6
Time Frame: 24 hours after surgery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
score on a scale | 2.0 [0 to 9] | 3 [0 to 7]

8. Secondary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Pain Scores
Description: as for outcome 6
Time Frame: 48 hours after surgery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
score on a scale | 2 [0 to 7] | 2 [0 to 7]

9. Secondary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Pain Scores
Description: as for outcome 6
Time Frame: 72 hours after surgery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
score on a scale | 2 [0 to 4] | 0.5 [0 to 7]

10. Secondary Outcome: Analgesic Effectiveness of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl as Measured by Change From Baseline in Patient Satisfaction With Recovery
Description: * Quality of Recovery -15 questionnaire
  * Part A has 10 questions that asks how the participant has been feeling in the last 24 hours with answers ranging from 0=none of the time to 10=all of the time
  * Part B has 5 questions asking the participant if they have had any of the following including pain, nausea, vomiting, anxiety, and depression) with answers ranging from 0=none of the time to 10=all of the time.
  * The total score allowed is 150 (range 0-150) with the higher the number the worse the participant is feeling and the lower the number the better the participant is feeling
Time Frame: At post operative day 2, discharge, and at 1-2 week follow-up
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 22 | 22
score on a scale
  Post-operative day 2 | -33 [-95 to 15] | -24 [-68 to 0]
  Discharge | -10 [-52 to 36] | -6 [-45 to 9]
  1-2 week follow-up | -18.5 [-59 to 37] | -10 [-41 to 8]

11. Secondary Outcome: Cost of Liposomal Bupivacaine (Exparel) Versus Bupivacaine HCl When Accounting for Length of Hospital Stay and Use of Other Analgesics
Time Frame: Up to 2 weeks post-operation
Population: Data was not collected for this outcome measure. There was no funding to collect or analyze the data. Also it was determined that the concept of cost was highly variable at the hospital and any data that was obtained would lack granular costs on most items. Lacking this granularity would make any results meaningless.
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were tracked from first administration of study drug until 30 days following the day of surgery.
Description: Only adverse events deemed to be serious, unexpected, severe, and related to the study drug will be recorded. Specifically, bleeding requiring blood transfusion, infection requiring readmission or surgery, life-threatening arrhythmias, would healing problems requiring surgical intervention, and reconstructive failures due to flap loss will be recorded and evaluated for relatedness.
Arm/Group | Group 1: Bupivicaine | Group 2: Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 8/22 | 10/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Bupivicaine (N=22) | Group 2: Liposomal Bupivacaine (N=22)
Failed Flap (Injury, poisoning and procedural complications) | 2 | 3
Wound dehiscence (abdomen requiring local debridement) (Injury, poisoning and procedural complications) | 4 | 1
Medical Flap Necrosis requiring debridement (Injury, poisoning and procedural complications) | 0 | 2
Flap Necrosis (Injury, poisoning and procedural complications) | 0 | 1
Flap hematoma requiring evacuation (Injury, poisoning and procedural complications) | 0 | 2
Breast reconstruction cellulitis (Infections and infestations) | 1 | 0
Abdominal wound cellulitis (Infections and infestations) | 0 | 1
Abdominal hematoma requiring evacauation (Injury, poisoning and procedural complications) | 0 | 1
Partial Flap Loss (Injury, poisoning and procedural complications) | 0 | 1
Late Flap Loss (Injury, poisoning and procedural complications) | 0 | 1
Delayed Pedicle TRAM Flap (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fascial dehiscence/hernia (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT02662036/Prot_SAP_000.pdf